CLINICAL TRIAL: NCT03673813
Title: Individual Nutritional Support at Home for Patients With Hypothalamic Obesity: Efficacy on Eating Behavior, Physical Activity, Physical Abilities, Weight Gain and Quality of Life
Brief Title: A Personalized Program of Physical Activity and Diet for Hypothalamic Obesity
Acronym: OH_APADIET
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: HAO17-Poitou_20170220; 2016-A00385-46 (Registry Identifier: RCB)
Record Dates: First submitted 2018-08-10; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-07

CONDITIONS: Hypothalamic Obesity
Keywords: Hypothalamic obesity; Prader-willi syndrome; Physical activity
MeSH Terms: conditions — Sexual Infantilism; Prader-Willi Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothalamic obesity (HO) is an obesity secondary to an alteration of the functioning of the hypothalamus, the central organ of energy homeostasis. The causes of OH are related to an hypothalamic lesion (eg craniopharyngioma) or to genetic diseases (ex: Prader-Willi syndrome). OH, which accounts for about 5 to 10% of obesity, is a complex handicap characterized by severe obesity associated with eating disorders, cognitive and behavioral disorders and sometimes a visual deficit, with a major impact on quality of life, morbidity and mortality. There is currently no specific treatment of HO. Management is essentially behavioral, based on daily support of eating behavior and physical activities (PA). OH is characterized by an intense and almost permanent hunger felt, a satiety disorder and an obsessive interest in food. The food education of the entourage is essential, the advise concern the control of the access to food and the setting up of a precise food frame on the quantities, with low energetic density, and schedules. OH is characterized by obesity with lean mass deficit. PA must therefore be regular, adapted to the disability and personalized to take into account cognitive deficits and behavioral disorders. Although the supervision of meals and daily PA is now recognized as fundamental in the care of these patients (National Program of Diagnosis and Care established by the French "Haute Autorité de Santé"), few studies have evaluated the effectiveness of programs with personalized support on global health. The investigators hypothesize that a personalized 4-month individual home-based counseling program on dietary counseling and PA can be effective to modify behaviors such as diet and PAs with an impact on changing weight and quality of life. The 16-week program includes a dietetic component (initial assessment with dietary care plan followed by a 30-minute telephone interview every month with dietician) and a PA component (two 1-hour individualized sessions, performed at home and supervised by a PA educator). Before and after the program, the investigators will evaluate habitual PA with an accelerometer, feeding behavior, physical functioning, weight change, body composition, quality of life and will constitute a biobank of serums, adipose tissues and stools. If the effectiveness of this program is demonstrated this will help to find ways to sustain this support by the institutions, to train professionals in the complex accompaniment of these patients. Finally this program set up as part of a rare disease can show the benefits in other populations of more common pathology (common severe obesity, intellectual disability, behavioral disorders).

DETAILED DESCRIPTION:
Hypothalamic obesity (HO) is defined as obesity secondary to impaired functioning of the hypothalamus nuclei, the central organ of energy and weight homeostasis. Among the causes of OH, there are those related to a hypothalamic lesion (lesional) such as craniopharyngioma (CP) or inflammatory (sarcoidosis, tuberculosis etc ..) and those called genetic, with gene abnormalities involved in the central regulation of energy homeostasis. The genetic causes of obesity can be either "monogenic" by mutation of genes involved in the leptin / melanocortin pathway, or "syndromic", defined by the association of obesity and other clinical signs (syndrome), such as Prader-Willi syndrome (PWS). PWS, which has a frequency of 1/15000 births, is one of the most well-known obesity-related syndromes. It is characterized by muscle hypotonia at birth, severe hyperphagia and dietary impulsivity, dysmorphic features, and intellectual disability with cognitive-behavioral abnormalities.

Although HO has various origins, it has a common phenotype with the presence of severe obesity, having a heavy impact on the morbidity and mortality. Obesity is multifactorial, associated with an increase in energy intake, a decrease in energy expenditure and an alteration of peripheral metabolism. First, impaired functioning of the hypothalamic nuclei leads to resistance to leptin and other hormones involved in the energy balance (GLP1, ghrelin etc.) leading to an increase in hunger and a lack of satiety responsible for hyperphagia. An alteration of the cognitive control of food intake and a hyper activation of the reward system have also been described in PWS, which can explain episodes of uncontrolled food impulsivity (food theft) and a high sensitivity to external stimuli in particular visualization of food. As such, it is a particularly interesting model for studying hyperphagia and alterations in the control of food intake. It should be noted that eating disorders vary from one individual to another but can also fluctuate for the same individual depending on the psychological state of the patients and their daily activities. The involvement of the autonomic nervous system leads to a decrease in the sympathetic tone responsible for a fall in resting energy expenditure. Indeed, there is a positive correlation between autonomic nervous system activity, basal metabolism, and spontaneous physical activity. In addition, endocrine deficits, present in HO, not or insufficiently substituted, such as gonadotropic, thyrotropic or somatotropic insufficiency have also a negative impact on resting energy expenditure. The total energy expenditure is also lowered by the low spontaneous physical activity (PA) of the patients in relation to the hypotonia described in these patients and a reduction of the spontaneous activation of the movements. In addition, sleep disorders (OSA, narcolepsy, daytime hypersomnolence) are common in patients with OH and may increase exercise fatiguability and difficulties for patients to do PA. Finally, visual disturbances (reduction of severe visual acuity by amputation of the visual field) associated with optic chiasm involvement in lesion-induced HO or induced by craniopharyngioma tumor resection, are also a limitation for PA and increase sedentary lifestyle. The absence of PA and the increase in sedentary lifestyle are associated with abnormal body composition with an increase in body fat at the expense of muscle mass . This is especially important in patients with PWS associated with developmental muscle hypotonia].

People with HO have often cognitive deficits, learning difficulties and social skills disorders. These are constant in the PWS but also in the lesional cause. All these factors lead to altering the quality of life. Thus, an impairment of quality of life has been demonstrated in 185 obese patients with craniopharyngioma in childhood. In our cohort of HO subjects, mood disorders assessed by the HAD score are common: 91% for lesional HO 50% for genetic HO and this is correlated with BMI. The Kendall-Taylor study shows that, in children with craniopharyngioma, the quality of life score depends on the age at diagnosis, the presence of somatotropic deficiency and BMI. At present, there is no specific treatment of HO. Drug treatments have been proposed such as melatonin, somatostatin analogue or sympathomimetics but with limited effects on weight and feeding behavior, resulting in no prescribing recommendations given the lack of randomized studies with sufficient patient samples. Sibutramine tested in patients with lesional or genetic HO, withdrawn from the market in France since 2010 for potentially deleterious effects on the cardiovascular system. GLP 1 analogues are also an interesting therapeutic approach in patients with craniopharyngioma with some efficacy on weight , but are currently reserved for diabetic patients. Regarding bariatric surgery, the HAS recommends that "the indication must be exceptional and discussed on a case by case basis". A meta-analysis of the results of bariatric surgery in 21 subjects with craniopharyngioma showed a weight loss at 1 year of 15.1 kg, in the same average as the obese general population operated. Nevertheless the subjects were selected (absence of important behavioral disorders) and the results concern only the short term. In genetic HO, especially PWS, the results of bariatric surgery should be used with caution. In terms of weight loss, the results are not as good, with medium-term weight regain, persistence of hyperphagia despite the reduction of the gastric pouch, and an increased risk of morbidity and mortality. Management is essentially behavioral, based on daily support of eating behavior and PA. Food management requires from a very young age for these patients, a permanent food control, to fight against primary impulsivity of central origin, can be a cause of frustration and behavioral disorders. Indeed, the genetic syndrome is characterized by intense and permanent hunger, a lack of satiety and an obsession for food. The affected patients are completely overwhelmed by this addictive behavior. It is extremely difficult or impossible for the child as for the adult with this syndrome to control his dietary intake. The entourage must therefore control access to food at home and abroad. This requires constant supervision. An early education of food in the family is essential because today it there is no possible and sustainable autonomy regarding diet for these patients. There is a strong need for coherence for caregivers to avoid unnecessary discussions and arguments. It is necessary to inform, prevent, associate the family and friendly entourage so that there is a coherence with the line of conduct chosen by all. Patients can not feel the signals that would allow them to have a meal like other people, so it is recommended to put in place a precise food frame on quantities and schedules, a low energy density food setting while providing sufficient food volume. A strict framework reassures and secures the patient because he has benchmarks. This is to reassure the person himself, to do everything possible to limit the temptations that are a source of tantrums and frustration. By respecting meal schedules and their composition ("food security"), by diverting patients' thinking, by occupying them, we can improve the food obsession of patients with HO. This specific and personalized dietary management is therefore necessary and essential. Physical activities are also a basic component of treating common obesity and its complications. It has a favorable effect on weight control, especially on the prevention of weight gain. In addition, PA has important beneficial effects on body composition. Regardless of weight loss, PA decreases total body fat and visceral abdominal fat. It also limits the loss of muscle mass during weight loss. Beyond its effects on weight control and body composition, PA is beneficially associated with many health parameters and decreases the risk of developing the major complications of obesity (type 2 diabetes and cardiovascular diseases). PA is also associated with an increase in quality of life. Finally, PA improves physical capacity that is often greatly diminished in obese subjects. Obesity is associated, on the one hand, with a decrease in cardiorespiratory fitness, muscular strength, functional capacity (observed for example during the 6-minute walk test) and, on the other hand, impaired balance and locomotion. Studies in patients with HO showed that patients had a low level of PA. Only one study measured PA level in the PWS. PA was measured using accelerometers in 28 young adults with moderate obesity. Only 25% of men and 15% of women achieved the minimum level of recommended PA and the average daily duration of moderate to high intensity AP was 14 minutes. Two studies measured PA level using accelerometers or pedometers in patients with craniopharyngioma. PA level was lower than that seen in normal weight subjects. In addition, the functional capacity of HO subjects appears to be impaired. For example, muscle strength, balance, and locomotion were assessed in 5 studies of 12 to 19 young adults with PWS and massive obesity. Muscle strength was significantly reduced compared to normal weight subjects, but also compared to control obese subjects. The balance was also altered, increasing the risk of falling. Finally, these patients adopted a different walking pattern (decreased walking speed and step length, increased double support time). Grolla et al. showed that a 4-week program, repeated 4 times a year, combining a low-calorie diet and a sustained program of PA (up to 7 hours of activities per day, such as walking, exercise bike , carpet exercises) reduced BMI of 2.5 kg / m2 and body fat by 2.5 kg in patients with PWS. Two other studies evaluated the effect of a PA program combining an initial stay of 2 weeks and a home-based training program for 6 months. During the initial 2 weeks, patients participated in 4 sessions per week, supervised by trained staff, during which they performed strength training and endurance exercises. During the following 6 months at home, patients autonomously performed 3 sessions per week of muscle strengthening. This program resulted in improved biomechanical parameters of the ankle and knee during walking. Other measured parameters (muscle strength, balance) were unchanged. Another study followed patients with PWS for 7 years during which patients regularly participated in rehabilitation programs combining PA, dietary management and physiotherapy. The results showed an improvement in the biomechanical parameters of gait. Thus, the management of HO should be comprehensive, residing in the control of the environmental risk factors of weight gain: management of hyperphagia by regular and personalized nutritional and dietary monitoring and appropriate medico-social support (educator, informed parents). Compulsive eating behavior can be reduced in a structured environment, with support and stimulation of other interests (especially physical activities and activities). In addition, a daily PA is essential to compensate for the decreased basic metabolism (see above). If support by PA and food management is now recognized as a fundamental element of the care of patients suffering from HO (National Program of Diagnosis and Care established by the HAS (Haute Autorité de Santé) http: // www.has-sante.fr/portail/upload/docs/application/pdf/2012-06/ald_hors_liste_-_pnds_on_the_syndrome_de_prader-willi.pdf), no study has evaluated the effectiveness of a personalized support program, framed and at home, focusing on dietary counseling, control of eating behavior and PA, on dietary behavior, patients' health status, physical activity volume and functional capacity, the evolution of weight and quality of life.

The hypothesis of the investigators is that a personalized home-based support program for dietary advice and PA for 4 months helps to change weight changes through behavioral changes such as increasing habitual physical activity, improving eating behavior, functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 to 60
* BMI ≥ 30kg / m² or MG ≥ 35% of total weight in men / 40% of total weight in women
* "Hypothalamic" obesity, defined as obesity with hyperphagia, and cognitive or neuropsychological disorders
* Entourage present (family or educator)
* Treatments not modified for at least 2 months (growth hormone, gonadotropic / thyrotropic / corticotropic substitution, Minirin, psychotropic drugs, etc.)
* Affiliation to a social security scheme

Exclusion Criteria:

* Introduction of new treatments in the 2 months preceding inclusion that can modify the feeding behavior (GLP1 analogues, Topiramate, psychotropic drugs, etc.).
* Decompensation of a cardiorespiratory or psychiatric pathology in the 3 months preceding the inclusion.
* Subject in a situation that, in the opinion of the investigator, could interfere with his / her optimal participation in the study (eg severe behavioral disorders) or constitute a particular risk for the patient (eg severe cardiorespiratory pathology).
* Contraindication to the physical activity discovered during the first evaluation (electrocardiogram abnormalities, abnormal stress test, abnormal cardiac echocardiography or effort scintigraphy, etc.).
* Subject in exclusion period after participation in another clinical trial.
* Pregnancy, breastfeeding.
* Interruption of more than 15 days of the foreseeable monitoring protocol (leave etc ..).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with hypothalamic obesity (lesional or genetic)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Compare the activity count (counts/mn) and pattern of activity (sedentarity time, light, moderate in %) measured objectively by an accelerometer before and after a 16-week program including a dietetic component and a PA component. Support over 4 months. | month 4
  PA volume indicator (taking into account the duration and intensity of the APs used) expressed in counts per minute, measured for 1 week objectively by an accelerometer (Actigraph GT3X®).advice and food intake control and a program of adapted physical activities at home in individual support.

SECONDARY OUTCOMES:
Measurement of weight in kg before and after the 4 months program | month 4
  In day hospital before and 4 months after supervised program (weight measured during the evaluations) and monthly measurement at home of the patient during 4 months (reported by the patient and his entourage and recorded by the dietician during the monthly telephone interview).
Evolution of the parameters evaluating the feeding behavior | month 4
  Score of Dyckens questionnaire ( 3 subscores behavior, drive and severity) before and after the 4 months program
Evolution the physical function before and after the 4 months program | month 4
  A 6-min walk test distance (meters)
Evolution of body composition (fat mass in kg and % evaluated by DEXA) | month 4
  lean mass and fat mass in kg and in% (DEXA)
Evolution of the quality of life | month 4
  self-questionnaire of the patient (SF12)